CLINICAL TRIAL: NCT03733457
Title: Technology-Assisted Stepped Care Intervention Pilot Study
Brief Title: Technology- Assisted Stepped Care Intervention Study
Acronym: TASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CIN001- {"TASC Intervention"}
Record Dates: First submitted 2018-10-30; First posted 2018-11-07 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TASC Intervention (Experimental): All participants receive Step 1 of the intervention. Participants who have adherence below or at 68% will step up to Step 2 or Step 3 after the third or fourth month in the study.
  Interventions: Behavioral: Technology-assisted Stepped-care

INTERVENTIONS:
Behavioral: Technology-assisted Stepped-care — Step 1 of the intervention includes educational materials related to asthma. Step 2 includes electronic monitoring of adherence and a text messaging intervention personally tailored to the participant. Step 3 includes problem solving telehealth sessions with a trained clinician.

SUMMARY:
The overall goal of this project is to demonstrate the feasibility, implementation, and preliminary efficacy of a technology-assisted stepped care (TASC) adherence-promotion intervention in adolescents with asthma. Preliminary efficacy will be demonstrated by improved adherence to daily inhaled corticosteroids as measured by Propeller Health electronic monitoring devices. The TASC intervention will result in improved disease severity measured by the Composite Asthma Severity Index (combining dose of asthma medication required, asthma symptom burden, and frequency of exacerbations and health care utilization) and lung function as measured by mobile spirometry. The TASC adherence-promotion intervention implementation will be successful as evidenced by high levels of feasibility (e.g., attendance), acceptability (20 item Acceptability Questionnaire), and usability (10 item Usability Scale).

DETAILED DESCRIPTION:
Up to thirty adolescents with asthma will be enrolled in an open label pilot trial of the TASC adherence-promotion intervention for a duration of five months. First, participants will complete baseline questionnaires related to demographic, and clinical predictors of adherence and asthma and a 4 week run-in phase to assess baseline adherence using electronic inhaler monitoring with a cellphone that is provided to them. Following the run-in period, all participants will receive Step 1 of the TASC intervention for a minimum of 4 weeks. Step 1 (Information) will include electronic educational information related to asthma symptoms and triggers, attacks, self-monitoring, treatments, action plans, and automated text message medication reminders. Following the initial four weeks of Step 1, adherence will be evaluated and a rate of less than 68% will serve as the cause for "stepping up" to the next level of the intervention. Adherence checks will continue to occur every four weeks for the duration of the study and adherence <68% will prompt movement from one level of treatment to the next. Participants may remain at a treatment level for more than four weeks and may complete 1, 2, or 3 interventions steps during the 5 month study depending on the adolescent's adherence. Step 2 (Motivation) will include electronic monitoring of adherence and personally tailored feedback via text messages. Adolescents will be given access to the adherence tracking smartphone app and graphs of their inhaler adherence. Adolescents will also receive brief, personalized text messages that provide supportive motivation and directive, tangible actions. Step 3 (Behavioral) will include problem-solving telehealth intervention with a trained clinician. Four telehealth sessions individually tailored to the unique needs and barriers of the adolescent will be provided. The primary outcome measure will be electronically-monitored adherence assessed at post-treatment. Secondary outcomes include asthma severity as well as process evaluation questions and quantitative measures of feasibility, acceptability, and satisfaction to demonstrate implementation.

ELIGIBILITY:
Inclusion Criteria:

* Patient age between 12-18 years
* Patient is diagnosed with severe-persistent or moderate-persistent asthma per NAEPP asthma guidelines
* Patient is prescribed at least one daily inhaled controller medication or a daily combination inhaled corticosteroid and long-acting beta-agonist and a beta-agonist bronchodilator
* English fluency for patient, caregiver, and clinician

Exclusion Criteria:

* Significant cognitive deficits that may interfere with comprehension per medical team or chart review.
* Diagnosis of serious mental illness (e.g., schizophrenia)
* Diagnosis of pervasive developmental disorder

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Electronic Monitoring | 5 Months
  The Propeller Health monitoring system includes a Bluetooth enabled sensor that attaches to the patient's inhaler. This sensor records every dose, or "puff", the patient takes and sends it to a corresponding online database that is accessible to study staff. Participants will be given this sensor at baseline.

SECONDARY OUTCOMES:
Composite Asthma Severity Index (CASI) | Baseline assessment and then once a month for 5 months
  The participants' composite asthma severity index score will be calculated through the TreatSmart program. TreatSmart will be used to determine the participant's symptom burden, health care utilization, systemic corticosteroid use, and current medication use to determine the level of asthma severity/control the participant has. The program also makes an initial treatment recommendation based on the National Asthma Education and Prevention Program (NAEPP asthma guidelines). Individuals are placed in Step 1 through Step 6 depending on the strength and frequency of their inhaled corticosteroid (1 being low dose and 6 being a high dose). In addition, individuals are categorized as very poorly controlled, not well controlled, or well controlled based on how frequently they have had asthma symptoms or used their rescue inhaler, gone to the hospital or urgent care, or received steroids for asthma symptoms.
Asthma Control Test (ACT) | Baseline assessment and then once a month for 5 months
  The ACT will be used as a measure of disease severity in this study. The ACT is a 5-question scoring tool designed for patients with asthma who are 12 years and older. The questions ask the patient to rate their asthma severity, symptom frequency, control, and inhaler use on a scale of 1-5. The total score is calculated by the sum of each response, which determines how well-controlled the patient's asthma is on a scale from 5-25.
Attendance/Participation rates | 5 months
  Participation rates will be measured 3 different ways. The first measure will be how often participants accessed the electronic material (educational materials and/or Propeller Health app), the second measure will be how many responses to directive text messaging were received, and the third measure will be attendance to the telehealth sessions.
Feasibility/Acceptability Questionnaire | 5 months
  A 5-31 item measure of format, content, length, skills and acceptability of the intervention will be given to participants in the form of a questionnaire at the end of each step and the end of the study. The feasibility section is on a scale of 0 to 4, 0 being the worst and 4 being the best. The acceptability questionnaire is on a scale from 'Not at all' to 'Very,' 'Not at all' being the worst and 'Very' being the best.
System Usability Scale | 5 months
  A 10 item, Likert scale giving a global view of usability will be given to participants in the form of a questionnaire at the end of each step and at the end of the study. The scale ranges from 'Strongly Disagree' to 'Strongly Agree, with half of the items reverse scored.
Treatment Fidelity | 5 months
  Treatment fidelity needed for the intervention will be assessed. Treatment fidelity will be assessed through fidelity checklists created specifically for each intervention session.
Time Needed for Intervention | 5 months
  Sessions will be timed and the number of weeks to complete the session will be tracked to determine the average length of time needed for the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Medical Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided